CLINICAL TRIAL: NCT04962412
Title: Predicting Poor Outcomes of Cardiac Surgery-Associated Acute Kidney Injury Using Novel Biomarkers
Status: Completed | Type: Observational
Sponsor: Guowei Tu (Other)
Responsible Party: Sponsor-Investigator, Guowei Tu, Scientific Secretary for Department of Critical Care Medcine, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Other Study IDs: B2021-390R
Record Dates: First submitted 2021-07-04; First posted 2021-07-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury; Critical Illness
Keywords: Acute kidney injury; Biomarker; AKI progression; Poor outcome; Furosemide Stress Test
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 365 Days
Biospecimen Retention: Samples Without DNA — Serial blood and urine samples for biomarker analysis were collected after surgery and then every 6 h in day 1 and then daily until discharge from ICU or for a maximum of 7 days, respectively. Plasma (EDTA), serum, and urine supernatants were frozen within 2 h of sample collection, stored at -80℃, and thawed immediately before analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Standard care "bundle" — The management for AKI patients were performed by implementing a standard care "bundle" suggested by the Kidney Disease Improving Global Outcome (KDIGO) guideline.

SUMMARY:
The aim of this study was to identify and validate novel biomarkers including functional tests for detecting AKI, AKI progression and other poor outcomes.

DETAILED DESCRIPTION:
Cardiac surgery-associated acute kidney injury (CSA-AKI) is the second most common type of AKI after septic AKI and is associated with increased mortality and morbidity. The progression of AKI with multiple organ failure can result in poor outcomes. Several novel biomarkers for earlier detection of AKI, discrimination of etiologies, and prediction of outcomes were developed. However, the availability of these novel biomarkers may be limited by its expense or reimbursement issues in different countries. In present study, we conduct a large cohort to identify and validate novel biomarkers including functional tests for detecting AKI, AKI progression and other poor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery were prospectively screened, and those who developed AKI within 48 hours post-surgery were included in the study.

Exclusion Criteria:

* History of End Stage Renal Disease or on Dialysis;
* prior kidney transplantation;
* patients with a DNR order;
* patients without written informed consent;
* pregnancy;
* moribund patients with expected death within 24 h or whose survival to 28 days was unlikely due to an uncontrollable comorbidity (i.e., end-stage liver or heart disease, untreatable malignancy)

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The incidence of cardiac surgery-associated AKI (CSA-AKI) varies from 5% to 42%. CSA-AKI is the second most common cause of AKI in the intensive care setting (after sepsis) and is independently associated with increased morbidity and mortality. Patients was diagnosed AKI by KDIGO criteria.
Sampling Method: Probability Sample
Enrollment: 3152 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
AKI progression | 7 days
  worsening of KDIGO stage within 1 week (progressing from stage 1 to either stage 2 or stage 3, or from stage 2 to stage 3).
  Patients diagnosed with progressive or persisting stage 3 AKI (stage 3 AKI for >3 consecutive days) were classified as having AKI progression.
  If patients who presented with stage 3 AKI but not requiring RRT subsequently required dialysis or developing persist severe AKI or death within 7 days, this was considered progression.

SECONDARY OUTCOMES:
Mortality | 365 days
  Mortality at 30 days, 90 days and 365 days
Receipt of renal replacement treatment | 365 days
  Patients received renal replacement treatment during hospital stay
Major adverse kidney events | 365 days
  MAKE was defined as the composite of≥25% loss in estimated glomerular filtration rate (eGFR), dialysis, or death. Estimated GFR was calculated from serum creatinine using the MDRD equation
Persistent AKI | 90 days
  Persistent AKI is characterized by the continuance of AKI by serum creatinine or urine output criteria (as defined by KDIGO) beyond 48h from AKI onset.
Persist severe AKI | 90 days
  Persistent severe AKI was defined as follows: Patients with stage 3 AKI at enrollment required a persistence of 72 hours or more to meet the end point.
  Patients enrolled at stage 2 AKI required a progression to stage 3 within 48 hours and a persistence at stage 3 for 72 consecutive hours to be considered end point positive.
  Additionally, patients with severe AKI who failed to achieve 72 hours due to death or the initiation of RRT were considered end point positive.
Length of stay in the ICU | 90 days
  Length of stay in the ICU
Length of stay in the hospital | 90 days
  Length of stay in the hospital
AKI progression to stage 3 | 7 days
  worsening of KDIGO stage to stage 3 within 1 week (progressing from stage 1 or stage 2 to stage 3).
AKI occurrence at 3 days | 3 days
  AKI was defined based on the Kidney Disease Improving Global Outcomes (KDIGO) criteria.
AKI occurrence at 7 days | 7 days
  AKI was defined based on the Kidney Disease Improving Global Outcomes (KDIGO) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, Professor, Study Director — Fudan University
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Su Y, Liu WJ, Zhao YF, Zhang YJ, Qiu Y, Lu ZH, Wang P, Lin S, Tu GW, Luo Z. Modified furosemide responsiveness index and biomarkers for AKI progression and prognosis: a prospective observational study. Ann Intensive Care. 2024 Oct 8;14(1):156. doi: 10.1186/s13613-024-01387-y. PMID 39379672